CLINICAL TRIAL: NCT01446523
Title: Serum Endotoxins, Inflammatory Mediators and MR Spectroscopy Before and After Treatment in Minimal Hepatic Encephalopathy
Brief Title: S. Endotoxin, Inflammatory Mediators and MRS Before and After Treatment in MHE
Acronym: endtxninHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Govind Ballabh Pant Hospital (Other Government)
Responsible Party: Principal Investigator, Barjesh Chander Sharma, Professor, Govind Ballabh Pant Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: endotoxins in MHE
Record Dates: First submitted 2011-09-11; First posted 2011-10-05 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Hepatic Encephalopathy
Keywords: endotoxins HE
MeSH Terms: conditions — Hepatic Encephalopathy | interventions — Lactulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactulose (Placebo Comparator): Group L receives lactulose Group NL receives placebo
  Interventions: Drug: Lactulose
- Placebo (Placebo Comparator): Group NL receives placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Syrup, 30 ml BD for 3 months in Gr. NL
  Arms: Placebo
Drug: Lactulose — Syrup 30 ml BD for 12 weeks
  Other Names: Duphalac , Looz
  Arms: Lactulose

SUMMARY:
The purpose of this study is to examine S.endotoxins , inflammatory mediators and Magnetic Resonance Spectroscopy (MRS) before and after treatment in patients of cirrhosis and minimal hepatic encephalopathy.

DETAILED DESCRIPTION:
60 patients of cirrhosis with Minimal Hepatic Encephalopathy (MHE) who fulfills the inclusion & exclusion criteria will be the part of study. Study patients will be divided in to two groups ( n=30 in each group).

Group L patients will receive lactulose therapy while Group NL will receive placebo. After 3 months , S.endotoxins , inflammatory mediators and MRS will be repeated in each group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Cirrhosis (Age 15 yr -70 yr )

Exclusion Criteria:

* Recent history of gastrointestinal bleed in last 6 weeks
* Active ongoing infection
* Creatinine >1.5mg%
* Electrolyte impairment. (S. Sodium < 130 meq/L, S. Potassium 3.5 meq/L or >5.0meq/L)
* H/O use of psychotropic drugs in last 6 weeks
* Recent alcohol use (< 6 week )
* H/O TIPS or shunt surgery.
* Hepatocellular Carcinoma
* Severe comorbidity as Congestive Heart Failure, Pulmonary disease, Neurological and Psychiatric problems impairing quality of life
* Poor vision precluding neuropsychological assessment

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Improvement of minimal hepatic encephalopathy | Baseline and at 12 weeks

SECONDARY OUTCOMES:
correlation between inflammatory mediators and grades of encephalopathy | Baseline and at 12 weeks
  To measure values of inflammatory mediators in different grades of encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Barjesh c Sharma, DM, Principal Investigator — GB Pant Hospital
Locations (1):
- BC Sharma, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Jain L, Sharma BC, Srivastava S, Puri SK, Sharma P, Sarin S. Serum endotoxin, inflammatory mediators, and magnetic resonance spectroscopy before and after treatment in patients with minimal hepatic encephalopathy. J Gastroenterol Hepatol. 2013 Jul;28(7):1187-93. doi: 10.1111/jgh.12160. PMID 23425082